CLINICAL TRIAL: NCT04899583
Title: A Prospective, Multicenter, Random Controlled Clinical Trail to Evaluate the Effectiveness and Safety of Sirolimus Coated Balloon Versus a Paclitaxel Coated Balloon in the Treatment of Coronary Bifurcation Lesion
Brief Title: ACOART SCB BIF: Treatment of Coronary Bifurcation Lesion by Sirolimus Coated Balloon vs Paclitaxel Coated Balloon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acotec Scientific Co., Ltd (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACOART SCB BIF
Record Dates: First submitted 2021-05-17; First posted 2021-05-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-05

CONDITIONS: Coronary Bifurcation Lesions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): a Sirolimus Coated Balloon
  Interventions: Device: Sirolimus Coated Balloon Catheter
- Control Group (Active Comparator): a Paclitaxel Coated Balloon Catheter
  Interventions: Device: a Paclitaxel Coated Balloon Catheter

INTERVENTIONS:
Device: Sirolimus Coated Balloon Catheter — a Sirolimus Coated Balloon Catheter designed and produced by Acotec
  Arms: Treatment Group
Device: a Paclitaxel Coated Balloon Catheter — a Paclitaxel Coated Balloon Catheter(trade name:Bingo)
  Arms: Control Group

SUMMARY:
The aim of this randomized controlled trial is to examine the treatment of coronary bifurcation lesion with a sirolimus coated balloon versus a paclitaxel coated balloon. This trial is designed as prospective, multicenter, randomized and open-label.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old
* Diagnosed as stable or unstable angina pectoris, asymptomatic myocardial ischemia or old myocardial infarction, or recent myocardial infarction in stable stage.
* Eligible for balloon dilatation or stent implantation.
* Subject (or legal guardian) understands the study requirements and procedures and provides written Informed Consent before any study tests or procedures are performed

Exclusion Criteria:

* AMI occurred within 7 days before operation
* The subjects had congestive heart failure or the heart function was classified as NYHA/KillipIV.
* Left ventricular ejection fraction (LVEF) < 35%
* History of heart transplantation
* The subjects had severe arrhythmias, such as high-risk ventricular extrasystole and / or ventricular tachycardia.
* The subjects had stroke, gastrointestinal bleeding or active ulcers, or had a high risk of bleeding in the past 6 months.
* Active bleeding physique or blood coagulation disorder
* Known renal insufficiency（eGFR<30ml/min）
* Contraindicated to anticoagulants or antiplatelet agents
* Has a history of percutaneous coronary intervention (PCI) within 6 months before enrollment.
* Has contraindications for coronary artery bypass grafting
* known to be allergic to aspirin, heparin, contrast agents, paclitaxel and sirolimus
* Life expectancy less than 12 months, or unable to complete a 12-month follow-up
* Pregnant or lactating females, or who plan to become pregnant during a follow-up period of 1 year after operation
* The subjects have participated in other drug property studies or device studies that have not yet completed the main end point.

Angiographic Inclusion Criteria:

* One target lesion (bifurcation lesion) in the coronary artery is allowed, and if there are coexistent non-bifurcated lesions requiring PCI intervention, only one lesion was accepted at most, and the target lesion should be treated after successful PCI treatment of non-target lesion.
* Target Lesion located in native coronary artery must be de novo
* Medina classification should be (1.1.1, 1.0.1, 0.1.1)
* Main branch of target lesion (%DS is ≥70% or ≥50% with clinical symptoms ) is suitable for stent implantation
* Target Lesion located in main branch should be covered by DES. Moreover, the residual stenosis ≤ 30%, TIMI flow is 3, no complications and branch vessel opening stenosis ≥ 70%.
* Reference vessel diameter of the branch is 2.0-4.0mm (by visual)
* Target lesion length ≤ 36mm (by visual)

Angiographic Exclusion Criteria:

* Target or non-target lesion located in left main
* Subjects who have non-target lesions of bifurcation
* The target lesion is trifurcation or multifurcation lesion.
* Main branch of target lesion located within 3 mm from the ostium of LAD or LCx or RCA
* The branch lesion is a diffuse long lesion, which could't covered by one DCB.
* Main or side branch is occlusive lesion, which TIMI flow is 0.
* Aneurysm existed in the blood vessel at the target lesion
* Side branch severely calcified or tortuous
* The blood pressure was too low to tolerate intracoronary injection of ≥ 100ug nitroglycerin
* Failure pre-dilatation of the side branch ostium (residual stenosis > 30% ,the blood flow in TIMI is not up to grade 3, or has dissection of type C or above according to NHLBI grade)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Diameter stenosis rate of bifurcation lesion determinated by Digital Substraction Angiography (DSA) at 9 months post procedure. | 9 months post procedure
  Defined as (1-minimum lumen diameter of target lesion/reference vessel diameter)*100% at 9 months post procedure.

SECONDARY OUTCOMES:
Rate of device success | Immediately after procedure
  Defined as the rate of successful delivery and withdrawal of the delivery catheter, and achieving a final in-lesion residual stenosis less than 30% and TIMI flow grade 3 by using the assigned device only.
Rate of lesion success | Immediately after procedure
  Defined as the rate of achieving a final in-lesion residual stenosis < 30% by visual estimate and TIMI flow grade 3 by using any percutaneous method.
Rate of procedure success | Immediately after procedure
  Defined as the rate of achieving lesion success without MACE (composite of cardiac death, MI and TLR events) .
Rate of target lesion failure (TLF) or device-related composite endpoints (DoCE） | 30 days, 6 months, 9 months, 12 months post procedure
  Defined as a composite rate of cardiac death, target vessel-related MI, or ischemia-driven TLR events at 30 days, 6 months, 9 months and 12 months post procedure.
Rate of patient-related composite endpoints (PoCE） | 30 days, 6 months, 9 months, 12 months post procedure
  Defined as a composite rate of all cause death, all cause-related MI or TLR events at 30 days, 6 months, 9 months and 12 months post procedure.
Diameter stenosis rate | 9 months post procedure
  Defined as the rate of restenosis (>50% diameter stenosis) of main vessel after 9 months at 9 months post procedure.
Late lumen loss (LLL) | 9 months post procedure
  Defined as the difference of minimum lumen diameter (MLD) from post procedure to 9 months follow-up, including late lumen loss of main vessel and side branch.
Angiographic binary restenosis (ABR) rate | 9 months post procedure
  Defined as the percentage rate of binary restenosis determined by angiographic at 9 months post procedure.
Rate of composite safety endpoint | 12 months post procedure
  Defined as a composite rate of all-cause death, cardiogenic death, myocardial infarction, target vessel-related myocardial infarction, incidence of thrombotic events (acute, subacute, late) defined by ARC at 12 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ge Junbo, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China